CLINICAL TRIAL: NCT04497181
Title: Study on the Effectiveness and Safety of Coil System for Intracranial Aneurysm Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I2017001223
Record Dates: First submitted 2020-07-26; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysms embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: Coil embolization surgery
- Control group (Sham Comparator)
  Interventions: Device: Coil embolization surgery

INTERVENTIONS:
Device: Coil embolization surgery — Embolization of aneurysms with various coils system

SUMMARY:
"Study on the effectiveness and safety of the coil system for the treatment of intracranial aneurysms embolization" was sponsored by Zhuhai Tongqiao Medical Technology Co., Ltd. The trial design is: prospective, multi-center, randomized, open, parallel positive control, and non-inferiority test. Purpose: To compare the data obtained by using the coil system produced by Zhuhai Tongqiao Medical Technology Co., Ltd. and the Axium Detachable Coil produced by Medtronic for the embolization of intracranial aneurysms to evaluate the effectiveness and safety of coil system for intracranial aneurysms embolization.

DETAILED DESCRIPTION:
"Study on the effectiveness and safety of the coil system for the treatment of intracranial aneurysms embolization" was sponsored by Zhuhai Tongqiao Medical Technology Co., Ltd. The team leader is Shanghai Changhai Hospital and the Second Affiliated Hospital of Zhejiang University School of Medicine. The trial design is: prospective, multi-center, randomized, open, parallel positive control, and non-inferiority test. Purpose: To compare the data obtained by using the coil system produced by Zhuhai Tongqiao Medical Technology Co., Ltd. and the Axium Detachable Coil produced by Medtronic for the embolization of intracranial aneurysms to evaluate the effectiveness and safety of coil system for intracranial aneurysms embolization. Sample: 228 cases. The subjects will be randomly assigned to the test group or the control group, with 114 cases in each group.

ELIGIBILITY:
Inclusion Criteria:

* An intracranial aneurysm was diagnosed by DSA examination of whole cerebral blood vessels, and it is planned to use a coil for the embolization of the target aneurysm
* The subject can understand the purpose of the research, show sufficient compliance with the research protocol, and sign an informed consent form

Exclusion Criteria:

* Multiple aneurysms
* Blood alveolar aneurysm, fusiform aneurysm, pseudoaneurysm, dissecting aneurysm, infectious aneurysm with arteriovenous malformation
* mRS score ≥ 3
* Hunt and Hess rating≥4
* Emergency ruptured aneurysms who need stent
* The target aneurysm has previously been treated with vascular embolization or surgery
* Patients with severe stenosis of the tumor-bearing artery
* PLT<60*10⁹ or INR>1.5
* Having vital organ failure or other serious diseases
* Received major surgery within 30 days before enrollment, or planned to undergo surgery within 90 days after enrollment
* History of allergy or contraindications to antiplatelet drugs, anticoagulant drugs, anesthetics, or contrast agents
* Patiens with a history of allergies to platinum and tungsten metals
* Life expectancy <12 months
* Pregnant or breastfeeding women
* Participated in other drug or device clinical trials within 1 month before signing the informed consent
* Other situations that the researcher judges are not suitable for inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Embolization success rate | 6 months
  Embolization success rate at 6-month after surgery

SECONDARY OUTCOMES:
Aneurysm recurrence rate | 6 months
  Aneurysm recurrence rate at 6-month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: jianmin zhang, M.D., Principal Investigator — Department of neurosurgery
Locations (1):
- Jianmin Zhang, Hangzhou, Zhejiang, China